CLINICAL TRIAL: NCT04017559
Title: Assessing the Clinical Impact of Motivational Interviewing on Inhaled Antibiotic Adherence in Cystic Fibrosis
Brief Title: Clinical Impact of MI on Inhaled Antibiotic Adherence in Cystic Fibrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 14074DD-AS
Record Dates: First submitted 2019-07-10; First posted 2019-07-12 (Actual); Last update posted 2019-07-12 (Actual); Status verified 2019-07

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention cohort (Experimental): All participants were entered into the intervention cohort to receive the Motivational Interviewing intervention
  Interventions: Behavioral: Motivational Interviewing

INTERVENTIONS:
Behavioral: Motivational Interviewing — A pharmacist trained in MI delivered three recorded MI sessions over 2 months, with follow up at 3, 4 and 6 months.

SUMMARY:
Adherence to treatment is a major challenge in cystic fibrosis (CF). Motivational Interviewing (MI) is increasingly used to address this, but its effectiveness is unknown. We investigated the clinical impact of an MI intervention, delivered by a specifically trained pharmacist, on adherence to inhaled antibiotics (IA).

DETAILED DESCRIPTION:
Adherence to treatment is a major challenge in cystic fibrosis (CF). Motivational Interviewing (MI) is increasingly used to address this, but its effectiveness is unknown. We investigated the clinical impact of an MI intervention, delivered by a specifically trained pharmacist, on adherence to inhaled antibiotics (IA).

Adults with CF were recruited through the Regional CF Centre. A pharmacist trained in MI delivered three recorded MI sessions over 2 months, with follow up at 3, 4 and 6 months. Demographics, ppFEV1, BMI, adherence (IA collection rates) and additional antibiotic use were collected during the study and for 6 months prior. Treatment Quality and Satisfaction (TQSM), self-reported adherence (Moriskey Medication Adherence Scale-8 (MMAS-8)), Quality Of Life (CF Questionnaire-Revised (CFQ-R)) and sputum Pseudomonas aeruginosa (Pa) density were assessed at each study visit. Statistical analysis compared outcomes pre and post-intervention and variation during the intervention period.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients with a documented diagnosis of CF aged ≥18 years on the date of informed consent
2. Known chronic infection with Pa, as defined by the Leeds criteria
3. Has been prescribed inhaled colomycin and/or tobramycin and/or aztreonam for a minimum of 3 months prior to study enrolment
4. Able to provide written informed consent
5. Able to understand and comply with protocol requirements and instructions
6. Has been identified by the physician during routine appointments as having difficulties with adherence to their inhaled therapies

Exclusion Criteria:

1. Patients that do not expectorate sputum spontaneously
2. Inability to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2014-10-22 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-05-17 (Actual)

PRIMARY OUTCOMES:
Inhaled Antibiotic collection percentage | 6 months preceding intervention compared to end of 6 month intervention period
  Change in adherence to Inhaled Antibiotic measured by collection from pharmacy in 6 months before intervention and at end of intervention

SECONDARY OUTCOMES:
Percent Predicted Forced Expiratory Volume in 1 second (ppFEV1) | 6 months
  Change in ppFEV1 from start of study to end of study (6 months)
Body Mass Index (BMI) | 6 months
  Change in BMI from start of study to end of study (6 months)
Need for additional Intra-venous or oral antibiotics | 6 months
  change in additional antibiotic days from 6 months preceding the intervention to end of intervention period
Treatment quality and satisfaction (TQSM) | 6 months
  Change in TQSM from start to end of intervention period
Self reported adherence using "Moriskey Medication Adherence 8" questionnaire (MMAS-8) | 6 months
  Change in MMAS-8 from start to end of intervention period
Density of Pseudomonas growth in sputum | 6 months
  Change in density of pseudomonas growth from start to end of intervention period
Quality of life measured by CFQ-R | 6 months
  Change in quality of life from start to end of intervention period

IPD SHARING:
Plan to Share IPD: No